CLINICAL TRIAL: NCT01038349
Title: Applications for Methotrexate Optimization in Rheumatoid Arthritis
Acronym: AMORA
Status: Completed | Type: Observational
Sponsor: Cypress Bioscience, Inc. (Industry)
Responsible Party: R. Michael Gendreau, M.D., Ph.D, Vice President, Chief Medical Officer, Cypress Bioscience, Inc
Other Study IDs: CYP-D-001
Record Dates: First submitted 2009-12-09; First posted 2009-12-23 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Avise PG - Diagnostic test — Eligible patients will receive an Avise PG test
  Other Names: Measure of methotrexate polyglutamates test

SUMMARY:
The goal of this study is to enable the study sponsor to assess the impact of a marketed or validated blood test has on physicians' clinical treatment decision making when treating RA patients who have been taking methotrexate.

Ultimately, the blood test will allow treating physicians to modify current methotrexate therapy in partially responding Rheumatoid Arthritis (RA) patients' therapy, on an individualized basis, as a means of improving clinical outcomes.

The study requires a blood sample from RA patients who have been on methotrexate therapy for a minimum of 3 months and are having an inadequate response to therapy. Physicians will then be provided with the results of the test indicating the methotrexate polyglutamate (active metabolites of methotrexate) levels in the patient's red blood cells as a means to help determine whether a patient's exposure to methotrexate has been optimized.

DETAILED DESCRIPTION:
This study is currently enrolling individuals who have an established diagnosis of RA and are receiving methotrexate as part of their therapy. Patients are required to submit a blood sample. There is no cost to volunteers who participate.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and sign the informed consent form
* Able to read, write, and speak English
* ≥18 years of age
* Diagnosed with RA within past 24 months (waiver)
* Taking oral methotrexate therapy for a minimum of 3 months
* Considered to have an insufficient response to methotrexate and therefore a candidate for change to therapy, including changing MTX dose or changing route of delivery, or adding or switching DMARDs (including but not limited to biologic DMARDs)

Exclusion Criteria:

* Prior exposure of the study center, study physician or study patient to the Avise PG laboratory test
* Patients with known abnormal hepatic and or hematological parameters
* Use of prednisone >10mg/day (or its equivalent)
* Rheumatologic diagnosis other than primary RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care and Rheumatology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To assess the impact of the Avise PG test on physician's clinical treatment decision making process when assessing RA patients having an inadequate response to current MTX therapy. | Outcome is determined following the receipt of Avise PG test result

CONTACTS AND LOCATIONS:
Overall Officials: R. Michael Gendreau, M.D., Ph.D., Study Director — Cypress Bioscience, Inc.